CLINICAL TRIAL: NCT07023705
Title: Monocyte To Large Platelet Ratio As A Diagnostic Marker For Acute Pulmonary Embolism
Brief Title: MLPR As A Diagnostic Marker For Acute Pulmonary Embolism
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Kheder Aly Awad, Assistant Lecturer, Ain Shams University
Other Study IDs: FMASU MLPR 286
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Pulmonary Embolism (Diagnosis); Diagnosis
MeSH Terms: conditions — Pulmonary Embolism; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pulmonary embolism: Group that is confirmed to have pulmonary embolism by positive CTPA finding filling defect.
  Interventions: Diagnostic Test: Monocyte to Large Platelet Ratio (MLPR)
- Non-Pulmonary embolism: Group that have pulmonary embolism diagnosis was excluded by negative CTPA finding.
  Interventions: Diagnostic Test: Monocyte to Large Platelet Ratio (MLPR)

INTERVENTIONS:
Diagnostic Test: Monocyte to Large Platelet Ratio (MLPR) — Admission laboratory values were used to calculate the Monocyte-to-Large Platelet Ratio (MLPR) by dividing the absolute monocyte count by the large platelet count. These values were obtained from blood samples collected before any treatment was administered.

SUMMARY:
A retrospective study to assess the utility of hematological marker (monocyte to large platelet ratio) to diagnose patients with pulmonary embolism

DETAILED DESCRIPTION:
The investigators conducted a retrospective review of emergency department records of patients who presented with signs and symptoms suggestive of pulmonary embolism (PE) and underwent CT pulmonary angiography (CTPA) for diagnosis. Hematological laboratory findings obtained prior to any treatment were collected and compared between two groups based on CTPA results: those with confirmed PE (CT positive) and those without PE (CT negative).

ELIGIBILITY:
Inclusion Criteria:

* Only patients with the results of full blood count and white blood cell differentiation, measured before the treatment of suspected PE.
* Patients underwent CT pulmonary angiography to confirm or exclude pulmonary embolism diagnosis.

Exclusion Criteria:

* Patient with history of any myeloproliferative disorder, myelofibrosis, Glanzmann thrombasthenia, May-Hegglin anomaly, Bernard-Soulier syndrome, suspicion of disseminated intravascular coagulation.
* Patient receiving any anticoagulant drug at a therapeutic dose.
* Patient with blood transfusion in the last 2 months.
* Patients with acute coronary syndrome, pulmonary edema.
* Patient on immunosuppressive drugs , Oral contraceptive pills .
* Patients with severe renal or hepatic disease.
* Patients with Stroke.
* Patients with malignancy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting to the emergency department with signs and symptoms of pulmonary embolism who underwent CT pulmonary angiography for diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Monocyte-to-Large Platelet Ratio (MLPR) | At emergency department admission (baseline lab measurement) before any treatment.
  A ratio between monocyte absolute count and the large platelets count (MLPR) values compared between groups using Mann-Whitney U test; diagnostic accuracy evaluated by area under the curve (AUC) , sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV).

SECONDARY OUTCOMES:
Mean platelet volume (MPV) | At emergency department admission (baseline lab measurement) before any treatment.
  MPV values compared between groups using Mann-Whitney U test; diagnostic accuracy evaluated by AUC, sensitivity, specificity, PPV, and NPV.
Neutrophil to Lymphocyte Ratio (NLR) | At emergency department admission (baseline lab measurement) before any treatment.
  The ratio between absolute neutrophil and absolute lymphocytes count (NLR) values compared between groups using Mann-Whitney U test; diagnostic accuracy evaluated by AUC, sensitivity, specificity, PPV, and NPV.
D-Dimer Levels | At emergency department admission (baseline lab measurement) before any treatment.
  D-Dimer concentration values compared between groups using Mann-Whitney U test; diagnostic accuracy evaluated by AUC, sensitivity, specificity, PPV, and NPV.
Platelet Distribution Width (PDW) | At emergency department admission (baseline lab measurement) before any treatment.
  PDW values compared between groups using Mann-Whitney U test; diagnostic accuracy evaluated by AUC, sensitivity, specificity, PPV, and NPV.
Platelet To Lymphocyte Ratio (PLR) | At emergency department admission (baseline lab measurement) before any treatment.
  The ratio between total platelets count and absolute lymphocytes count (PLR) values compared between groups using Mann-Whitney U test; diagnostic accuracy evaluated by AUC, sensitivity, specificity, PPV, and NPV.

CONTACTS AND LOCATIONS:
Overall Officials: Reem H Elkabarity, Professor, Study Chair — Ain Shams University; Hadil M Abdelhamid, Professor, Study Director — Ain Shams University; Azza Lotfy, Professor, Study Director — Ain Shams University; Mohamed k Awad, Lecturer, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Granger V, Faille D, Marani V, Noel B, Gallais Y, Szely N, Flament H, Pallardy M, Chollet-Martin S, de Chaisemartin L. Human blood monocytes are able to form extracellular traps. J Leukoc Biol. 2017 Sep;102(3):775-781. doi: 10.1189/jlb.3MA0916-411R. Epub 2017 May 2. PMID 28465447
- [Background] Moharamzadeh P, Rahmani F, Foroughifar S, Shahsavarinia K. Reliability of Platelet Indices for Diagnosing Pulmonary Embolism; a Brief Report. Adv J Emerg Med. 2019 Apr 28;3(3):e27. doi: 10.22114/ajem.v0i0.137. eCollection 2019 Summer. PMID 31410404
- [Background] Talay F, Ocak T, Alcelik A, Erkuran K, Akkaya A, Duran A, Demirhan A, Kar Kurt O, Asuk Z. A new diagnostic marker for acute pulmonary embolism in emergency department: mean platelet volume. Afr Health Sci. 2014 Mar;14(1):94-9. doi: 10.4314/ahs.v14i1.15. PMID 26060464
- [Result] Bialas AJ, Kornicki K, Ciebiada M, Antczak A, Sitarek P, Milkowska-Dymanowska J, Piotrowski WJ, Gorski P. Monocyte to large platelet ratio as a diagnostic tool for pulmonary embolism in patients with acute exacerbation of chronic obstructive pulmonary disease. Pol Arch Intern Med. 2018 Jan 31;128(1):15-23. doi: 10.20452/pamw.4141. Epub 2017 Nov 7. PMID 29112185